CLINICAL TRIAL: NCT01043055
Title: Evaluation the Diagnostic Ability of the CDT to Detect Breast Cancer Among Women Population Over Age 40
Brief Title: Evaluation the Diagnostic Ability of the Cancer Detection Technology (CDT) to Detect Breast Cancer Among Women Population Over Age 40
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Tamar Peretz, Head of Oncology Department, Hadassah Medical Organization
Other Study IDs: 044809-HMO-CTIL
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast Cancer Patients
- Healthy Control Group

SUMMARY:
This study aimed to validate the diagnostic ability of the CDT (cancer detection technology) software to detect breast cancer among women population.

DETAILED DESCRIPTION:
Breast cancer diagnosis is a rapidly expanding research field, whose early-stage detection may reduce the burden of the disease and permit more effective treatment. It is well documented that tumor growth requires specific conditions for its development from the occurrence of a mutation to a clinically detectable cancer. It has been shown that living peripheral blood mononuclear cells (PBMC) have different ability of cytosolic enzymes (esterases) to convert hydrophobic substrate fluorescein diacetate (FDA) into hydrophilic fluorescent fluorescein. It depends on PBMC cycle stage, size, surface state, physiological states, such as activation and apoptosis.

The important step of breast cancer genesis is the early change of functional activity of cytosolic enzymes (esterases) in peripheral blood mononuclear cells. Such transformations in PBMC may be detected accurately by an existing device Flowcytometer (FACS™ MultiSET™ System, company "Becton Dickinson" GmbH, USA), where measurements of fluorescence polarization and enzymatic hydrolysis of FDA substrate are recorded. A conclusion about presentation of breast cancer among examined women is achieved by "CDT" (cancer detection technology) software, which analyzes mathematically the results of fluorescence polarization and enzymatic hydrolysis.

Moreover, the combined biochemical model together with additional prognostic parameters (such as age, ethnic group, gynecological and obstetric anamnesis) increases the validity (accuracy, sensitivity and specificity) of the diagnostic conclusion.

Diagnostic Solution of the CDT:

1. Mathematical processing of specific blood analysis in device Flowcytometer.
2. Mathematical evaluation of specific prognostic parameters

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Breast Cancer Patients for Experimental Group:

1. Patient is over the age of 40.
2. Patient is willing to participate as evidenced by signing the written informed consent form.
3. Patient referred to the Department of Oncology/ Surgery for operative treatment of breast cancer with previously detected disease. Positive conventional tests finding can include (but not limited to) the record of screening or diagnostic mammography, blood oncomarkers, breast ultrasound, breast CT, biopsy.
4. Non-treated patients (w/o previous chemotherapy, hormonal drugs and radiotherapy).
5. Patient without other cancer locations

Inclusion Criteria for Presumably Healthy Subjects for Control Group:

1. Subjects over the age of 40.
2. Subjects who are willing to participate as evidenced by signing the written informed consent form.
3. Subjects who are presumably healthy and without breast pathologies' symptoms and family history of breast cancer, i.e., breast disease (except history of functional breast problems, e.g., mastitis within lactation period) has been ruled out based on physician anamnesis
4. Subjects with negative results of screening mammography.
5. Subjects without taking of any hormonal medicines

Exclusion Criteria:

1. Subjects with any known cancer in other internal organs or systems.
2. Subjects with high fever presentation (more than 38.5).
3. Subjects with known breast disease undergoing treatment for the disease.
4. Pregnant or lactating women

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients over age 40 before treatment. Healthy women recruited in Check Up institute from asymptomatic women over age 40, referred to screening mammography and received the negative result of mammography.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
To validate the diagnostic ability of the CDT to detect breast cancer among women population over age 40 | one year

SECONDARY OUTCOMES:
To correlate the technology with standard test - screening mammography and biopsy | two years
To validate and compare the diagnostic ability of the CDT for detection of breast cancer | two years

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Peretz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Jerusalem, Israel